CLINICAL TRIAL: NCT04942626
Title: Capecitabine-based Chemoradiotherapy in Combination With the IL-1 Receptor Antagonist Anakinra for Rectal Cancer Patients. A Phase I Trial of the German Rectal Cancer Study Group
Brief Title: Capecitabine-based Chemoradiotherapy in Combination With the IL-1 Receptor Antagonist Anakinra for Rectal Cancer Patients
Acronym: ACO/ARO/AIO-21
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Claus Rödel, Prof. Dr. med. Dr., Clinical Chair, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACO/ARO/AIO-21
Record Dates: First submitted 2021-05-25; First posted 2021-06-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Interleukin 1 Receptor Antagonist Protein; Capecitabine; Radiotherapy; Receptors, CCR

STUDY DESIGN:
Intervention Model Description: 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiotherapy with Anakinra followed by either TME surgery or Watch and Wait (Other): Capecitabine 500 mg/m2 bid or Capecitabine 650 mg/m2 bid or Capecitabine 825 mg/m2 bid combined with Radiotherapy and Kineret
  Interventions: Drug: Kineret 100 MG in 0.67 ML Prefilled Syringe; Drug: Capecitabine; Radiation: Radiotherapy; Procedure: Watch and Wait (cCR) or TME surgery (non-cCR)

INTERVENTIONS:
Drug: Kineret 100 MG in 0.67 ML Prefilled Syringe — Anakinra 100 mg s.c. (Kineret) will be administered from day -10 (i.e. 10 days before initiation of RT) to the last day of RT.
Drug: Capecitabine — Capecitabine will be administered using a 3+3 dose escalation design (500 mg/m2 bid, 650 mg/m2 bid and 825 mg/m2 bid po, respectively) from day 1 to day 40 of RT including weekends.
Radiation: Radiotherapy — PTV: 1.8 Gy to 45 Gy (#28 fractions) to the primary tumor and pelvic lymph nodes; followed by a sequential boost of 1.8 Gy to 9 Gy (#5 fractions) to the gross tumor volume
Procedure: Watch and Wait (cCR) or TME surgery (non-cCR) — Restaging to evaluate tumor response will be conducted 10 weeks after completion of CRT. For patients achieving a clinical complete response (cCR), a Watch and Wait (W&W) option with close follow-up is scheduled. In case of non-cCR, immediate total mesorectal excision (TME) surgery is recommended. According to the current German S3-guidelines, adjuvant chemotherapy is optional.
  Other Names: W&W or TME

SUMMARY:
The ACO/ARO/AIO-21 investigator-driven, open-labeled, phase I drug re-purposing trial will assess whether the IL-1 receptor antagonist Anakinra can be safely combined with fluoropyrimidine-based chemoradiotherapy (CRT) in patients with rectal cancer.

DETAILED DESCRIPTION:
Preoperative fluoropyrimidine-based chemoradiotherapy (CRT) and total mesorectal excision (TME) surgery 6-10 weeks thereafter, followed by optional adjuvant chemotherapy, has been the standard multimodal treatment for patients with UICC stage II and III rectal cancer during the last two decades. With this, pathological complete response rates (pCR) are in the range of 10%, 3 year-local failure rates in the range of 5%, distant recurrences occur in 25-30% of patients, and 3 years disease-free survival (DFS) amounts to 70%. More recently, total neoadjuvant treatment (TNT) with either 5x5 Gy or fluoropyrimidine-CRT, followed by consolidation chemotherapy with fluorouracil (or capecitabine) and oxaliplatin (FOLFOX/CAPOX), and TME, has significantly improved pCR and DFS compared to standard preoperative FU-CRT (+/- adjuvant chemotherapy) in recent phase 3 trials for patients with high-risk rectal cancer and has recently been accepted as standard treatment for this patient subgroup. In contrast, it remains unclear whether patients with intermediate risk rectal cancer benefit from TNT (currently under investigation in trials), whereas elderly and frail patients are not eligible for TNT and are rather be treated with 5x5 Gy or capecitabine-CRT alone. IL-1 is an inflammatory cytokine that plays a key role in tumor formation, progression and therapy resistance. Extensive studies of our group have showed that IL-1 mediates CRT resistance and disease progression in rectal cancer. Thus, blockade of IL-1 signaling using Anakinra constitutes an attractive option to significantly improve prognosis. The ACO/ARO/AIO-21 phase I drug re-purposing trial will assess whether the IL-1RA Anakinra can be safely combined with CRT in patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with histologically confirmed diagnosis of rectal adenocarcinoma localized 0 - 12 cm from the anocutaneous line as measured by rigid rectoscopy (i.e. lower and middle third of the rectum)
* Staging requirements: High-resolution, thin-sliced (i.e. 3 mm) magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
* Patients with MRI-defined low risk rectal cancer with the presence of at least one of the following conditions:

  * cT2N0 or cT3a/bN0 tumors ≤6 cm from the anocutaneous line that would require abdominoperineal resection or permanent colostomy
  * Any rectal cancer of the upper third (12-16 cm) requiring FU-CRT according to German S3 guideline recommendations (i.e. cT4, mrCRM+, extensive N+)
* Patients with MRI-defined intermediate/high risk rectal cancer, but not eligible for TNT (oxaliplatin-containing) protocols:

  * any cT3 if the distal extent of the tumor is < 6 cm from the anocutaneous line, or
  * cT3c/d in the middle third of the rectum (≥ 6-12 cm) with MRI evidence of extramural tumor spread into the mesorectal fat of more than 5 mm (>cT3b), or
  * cT3 with clear cN1 based on strict MRI-criteria (see appendix)
  * cT4 tumors, or
  * Tany middle/low third of rectum with clear MRI criteria for N2
  * mrCRM+ (≤ 1mm), or
  * Extramural venous invasion (EMVI+)
* Trans-rectal endoscopic ultrasound (EUS) is additionally used when MRI is not definitive to exclude early cT1 disease in the lower third or middle third of the rectum.
* Spiral-CT of the abdomen and chest to exclude distant metastases.
* Aged at least 18 years. No upper age limit
* WHO/ECOG Performance Status ≤1
* Adequate hematological, hepatic, renal and metabolic function parameters:

  * Leukocytes ≥ 3.000/mm^3, ANC ≥ 1.500/mm^3, platelets ≥ 100.000/mm^3, Hb > 9 g/dl
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * Bilirubin ≤ 2.0 mg/dl, SGOT-SGPT, and AP ≤ 3 x upper limit of normal
* Informed consent of the patient

Exclusion Criteria:

* Distant metastases (to be excluded by CT scan of the thorax and abdomen)
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Major surgery within the last 4 weeks prior to inclusion
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception during treatment and for 6 months after the end of treatment.
* On-treatment participation in a clinical study in the period 30 days prior to inclusion
* Previous or current drug abuse
* Other concomitant antineoplastic therapy
* Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active, uncontrolled infections, active, disseminated coagulation disorder
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrolment
* Prior or concurrent malignancy ≤ 3 years prior to enrolment in study (Exception: non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1), if the patient is continuously disease-free
* Known allergic reactions on study medication
* Known dihydropyrimidine dehydrogenase deficiency
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial).
* History of severe hepatic impairment (e.g. Child-Pugh = Grade C)
* Moderate (Creatinine Clearance 30 to 49 mL/minute), severe (Creatinine Clearance <30 mL/minute) renal impairment
* Neutropenia (neutrophil count <1.5x109/l)
* Known hypersensitivity to Anakinra or E. coli derived proteins, Anakinra or any of the components of the product
* Asthma
* Patients with clinically significant bacterial, fungal, parasitic or viral infection, which require acute therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed
* Patients with known active hepatitis B, C or who are HIV-positive or who are at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Prior test results obtained as part of standard of care that confirm a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility and tests do not need to be repeated. Subjects with prior positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
* Subjects who are already using the following medications will not be allowed:

  * Tumor necrosis alpha inhibitors: Use on any of these biologics within 8 weeks of screening or baseline visit.
  * IL-6 inhibitors: Use of any IL-6 inhibitors within 8 weeks of screening or baseline visit
  * Janus Kinase inhibitors: Use of baricitinib, tofacinitib, upadacitinib, and ruxolitinib, oclacitinib, fedratinib, within 2 weeks from screening or baseline visit.
  * Bruton's tyrosine kinase inhibitors: Ibrutinib, acalabrutinib, zanubrutinib
  * CCR5 antagonist (CCR5 = C-C Chemokine Receptor Type 5; DMARD = Disease Modifying Anti-Rheumatic Drug): Leronlimab is also an immunomodulator.
  * DMARDs: cyclosporine, cyclophosphamide, mycophenolic acid, chlorambucil, penicillamine, azathioprine: Use within 6 months prior to screening or baseline visit.
  * Rituximab: Use of rituximab within 1 year of screening or baseline visit.
  * Abatacept: Use of abatacept within 8 weeks of screening or baseline visit.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
* Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 30 days (incl. live attenuated vaccine) of screening or 5 half-lives (whichever is longer) prior to the first dose of investigational product
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed
* History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or that might affect interpretation of the results of this study, or render the subject at high risk for treatment complications.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of safety for capecitabine administered concomitantly with standard radiotherapy in combination with Anakinra at a fixed dose of 100 mg s.c. | 16 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Identification of the maximum tolerated dose for capecitabine administered concomitantly with standard radiotherapy in combination with Anakinra at a fixed dose of 100 mg s.c | 16 weeks
  Identification of the maximum tolerated dose for capecitabine in combination with radiotherapy and Anakinra based on 3+3 design

SECONDARY OUTCOMES:
Postoperative complications of (salvage) surgery | 1 year
  Postoperative complications of (salvage) surgery
Late toxicity assessment according to NCI CTCAE V.5.0 | 3 years
  Late toxicity assessment according to NCI CTCAE V.5.0
Rate of W&W with or without local regrowth | 3 years
  Rate of W&W with or without local regrowth
Cumulative incidence of locoregional regrowth after cCR | 3 years
  cumulative incidence of locoregional regrowth after cCR
Rate of salvage surgery (LE/TME with or without APR/stoma) after locoregional regrowth | 3 years
  Rate of salvage surgery (LE/TME with or without APR/stoma) after locoregional regrowth
Cumulative incidence of local recurrence after (salvage) surgery | 3 years
  Cumulative incidence of local recurrence after (salvage) surgery
Cumulative incidence of distant recurrences | 3 years
  Cumulative incidence of distant recurrences
Disease-free survival | 3 years
  Disease-free survival
Overall survival | 3 years
  Overall survival
Pathological TNM-staging | 3 years
  Pathological TNM-staging based on TNM Classification of Malignant Tumors, 8th edition
R0 resection rate; | 3 years
  Rate of complete resection (R0)
negative circumferential resection rate | 3 years
  negative circumferential resection rate
Tumor regression grading according to Dworak | 3 years
  Tumor regression grading according to Dworak
Quality of TME according to MERCURY | 3 years
  Pathological tumor evaluations according to MERCURY classification
Quality of life based on treatment arm and surgical procedures/organ preservation | 3 years
  Quality of life based on EORTC-QLQs-C30
functional outcome based on treatment arm and surgical procedures/organ preservation | 3 years
  functional outcome based on Wexner score
Quality of life based on treatment arm and surgical procedures/organ preservation | 3 years
  Quality of life based on EORTC-QLQs-CR29
Quality of life based on treatment arm and surgical procedures/organ preservation | 3 years
  Quality of life based on EORTC-QLQs-CPIN20

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roedel, Prof. MD, Study Chair — University Hospital Goethe University Frankfurt
Locations (1):
- University Hospital Goethe University Frankfurt, Frankfurt, Germany